CLINICAL TRIAL: NCT05303155
Title: The Association of Gut Microbiota With Early Infection Stages of COVID-19 in Children
Brief Title: The Association of Gut Microbiota With COVID 19 Infection in Children
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hallym University Kangnam Sacred Heart Hospital (Other)
Responsible Party: Principal Investigator, Ky Young Cho, M.D., Ph.D., Hallym University Kangnam Sacred Heart Hospital
Other Study IDs: Covid 19 and Gut Microbiota
Record Dates: First submitted 2022-03-18; First posted 2022-03-31 (Actual); Last update posted 2023-05-19 (Actual); Status verified 2023-05

CONDITIONS: Coronavirus Infections; Gut Microbiome; Childhood ALL
MeSH Terms: conditions — Coronavirus Infections; Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Fecal microbiome
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient with COVID 19: Pediatric patient infected by COVID 19
  Interventions: Diagnostic Test: 16S rRNA sequencing
- Pediatric patient without infection of COVID 19: Pediatric patient without infection of COVID 19
  Interventions: Diagnostic Test: 16S rRNA sequencing

INTERVENTIONS:
Diagnostic Test: 16S rRNA sequencing — Fecal microbiome analysis using 16S rRNA sequencing

SUMMARY:
Although COVID-19 infects gastrointestinal tissues, little is known about the roles of gut commensal microbes in susceptibility to and severity of infection. The investigators will analyze the alterations in fecal microbiomes of patients with COVID-19 infection during hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* patients infected with COVID 19

Exclusion Criteria:

* congenital heart, renal, intestinal disease
* malignancy
* immunologic disease

Ages: 3 Months to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Those who were hospitalized because of the COVID 19 were enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2022-04-14 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
The analysis of fecal microbiome of patient with COVID 19 | through study completion, an average of 1 year
  The analysis of fecal microbiome of patient with COVID 19, using 16S rRNA sequencing

CONTACTS AND LOCATIONS:
Overall Officials: KY YOUNG CHO, MD, PhD, Principal Investigator — Hallym University Kangnam Sacred Heart Hospital
Locations (1):
- Hallym University Kangnam Sacred Heart Hospital, Seoul, South Korea